CLINICAL TRIAL: NCT02740426
Title: Peking University First Hospital
Brief Title: Prophylactic Intravesical Chemotherapy to Prevent Bladder Recurrence After Diagnostic Ureteroscopy for Primary Upper Tract Urothelial Carcinoma Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Xuesong Li, Director, Peking University First Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IUPU-16-UTUC
Record Dates: First submitted 2016-04-12; First posted 2016-04-15 (Estimated); Last update posted 2017-09-21 (Actual); Status verified 2017-09

CONDITIONS: Upper Tract Urothelial Carcinoma; Bladder Recurrence
MeSH Terms: interventions — pirarubicin

ARMS (2):
- Blank control (No Intervention): do not use prophylactic intravesical chemotherapy.
- Single intravesical instillation (Experimental): intravesical instillation within 24 hours postoperatively
  Interventions: Drug: Pirarubicin

INTERVENTIONS:
Drug: Pirarubicin — single immediate intravesical dose of pirarubicin (THP) intravesical therapy (THP 40 mg for 30 min) within 24 hours of ureteroscopy.
  Arms: Single intravesical instillation

SUMMARY:
This clinical trial is designed to evaluate the efficacy of single immediate intravesical chemotherapy instillation in the prevention of bladder recurrence after diagnostic ureteroscopy for upper tract urothelial carcinoma (UTUC) patients.

DETAILED DESCRIPTION:
INTRODUCTION

Upper tract urothelial carcinomas (UTUC) are relatively uncommon compared to bladder cancer and account for only 5-10% of urothelial carcinomas [Munoz et al., 2000; Siegel et al., 2012; Rouprêt et al. 2015], with an estimated annual incidence in Western countries of ~2 cases per 100,000 inhabitants. In 17% of cases, concurrent bladder cancer is present [Cosentino et al., 2013].

Urinary cytology, cystoscopy and computed tomograpy urography should be performed as the standard diagnostic work-up with the grade A of recommendation [Rouprêt et al., 2015]. Diagnostic ureteroscopy and biopsy should be performed, certainly in cases where additional information will impact treatment decisions. Such ureteroscopic biopsies can determine tumour grade in 90% of cases with a low false-negative rate [Rojas et al., 2012]. Ureteroscopy can prove invaluable in cases of suspected UTUC, especially when the diagnosis is equivocal, or if nephron sparing surgery is considered. However, it can pose potential hindrances, including difficulty in obtaining adequate tissue, inconsistent pathologic interpretation and prediction, and a high rate of upgrading and upstaging at the time of nephroureterectomy [Potretzke et al., 2015].

Recurrence in the bladder after management of UTUC occurs in 22-47% of UTUC patients [Xylinas et al., 2012; Zigeuner et al., 2006; Novara et al., 2008], compared with 2-6% in the contralateral upper tract [Li et al., 2010; Novara et al., 2009]. At our institution, we reported that 30.8% of UTUC patients developed intravesical recurrence, which was in line with the global trend [Fang et al., 2013]. Although the risk factors for development of bladder tumor post surgical management of UTUC were previously studied, considerable variations were observed in the literature. In previously published studies, we pointed out that lower tumor grade, tumor multifocality, concomitant carcinoma in situ (CIS), tumors located in the lower ureter, ureteroscopy history and unmethylated promoter of GDF15 and RASSF1A promoters were considered as predictors to develop bladder recurrence after surgery by univariate and multivariate analysis [Fang et al., 2013, Xiong et al., 2015]. As an effective tool to evaluate UTUCs visually or by biopsy, ureteroscopy was selectively used in early UTUC patients without atypical radiography. It was our hypothesis that retrograde flow, increased urine flow rate and intraluminal pressure might lead to the shedding of tumor cells (intraluminal tumor seeding is thought to contribute to intravesical recurrence after nephroureterectomy), which implant in the bladder to develop recurrences [Xiong et al., 2015].

AIM OF THE WORK This clinical trial is designed to evaluate the efficacy of single immediate intravesical chemotherapy instillation in the prevention of bladder recurrence after diagnostic ureteroscopy for UTUCs.

ELIGIBILITY:
Inclusion Criteria:

* Suspected UTUC patients without history of bladder tumor.
* Suspected UTUC patients without synchronous bladder tumor.
* Suspected UTUC patients without contralateral UTUCs.

Exclusion Criteria:

* Patients with history of bladder tumor.
* Patients with synchronous bladder tumor.
* Patients with contralateral UTUCs.
* Patients with advanced stage (T4).
* Patients with other malignant tumors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2016-08; Primary Completion 2021-05 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
intravesical recurrence-free survival | three years after surgery

SECONDARY OUTCOMES:
cancer-specific survival | three years after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China